CLINICAL TRIAL: NCT03378791
Title: Iron Bisglycinate Chelate or Ferrous Fumarate in Treatment of Iron Deficiency Anemia in Pregnant Women
Brief Title: Efficacy of Iron Bisglycinate in Treatment of Iron Deficiency Anemia in Pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS/15.10.05
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Iron Deficiency Anemia of Pregnancy
MeSH Terms: interventions — ferrous fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Group A (Experimental): Iron bisglycinate (27mg of elemental iron)
  Interventions: Drug: Iron bisglycinate Oral Tablet
- Group B (Active Comparator): Ferrous fumarate (115mg of elemental iron)
  Interventions: Drug: Ferrous Fumarate Oral Tablet

INTERVENTIONS:
Drug: Iron bisglycinate Oral Tablet
  Arms: Group A
Drug: Ferrous Fumarate Oral Tablet
  Arms: Group B

SUMMARY:
Anemia in pregnancy is defined by the World Health Organization as hemoglobin levels of ≤ 11 g/dl. Globally, a prevalence rate of 38% was estimated by the World Health Organization for pregnant women.Treatment of iron deficiency anemia during pregnancy remains a main public health issue. Oral iron salts have been recommended for treatment of iron deficiency anemia e.g. ferrous fumarate. Increasing the dose of ferrous fumarate will subsequently increase the bioavailability of iron preparation, however it also increases the frequency of gastrointestinal tract side effects e.g. nausea, constipation, diarrhea, flatulence, and black stained stools. Besides, the increased bioavailable ferrous fumarate may decrease by many foods and / or chelating drugs in the gastrointestinal tract which interfere with its absorption leading to variability in the hemoglobin correction during the treatment.

Ferrous bisglycinate is an iron amino acid chelate. It is formed by reaction of ferrous iron with two molecules of the amino acid glycine by a covalent bound in a process called chelation. Ferrous bisglycinate is claimed to have better patient compliance because of fewer gastrointestinal tract side effects. It is also claimed that ferrous bisglycinate improves iron absorption, storage and increase hemoglobin level better than the conventionally used iron salts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 20 to 40 years,
* 14-27 gestational weeks calculated from the first day of their last menstrual period and confirmed by ultrasound
* Singleton fetus
* hemoglobin level from 7-9.9 g/dL.

Exclusion Criteria:

* All women with high risk pregnancy e.g. hypertension, diabetes
* multiple pregnancy
* women with severe anemia (Hb >7 g/dl)
* anemia due to other causes than iron deficiency as chronic blood loss, hemolytic anemia or thalassemia.
* women with hepatic, renal or cardiovascular abnormality; women with peptic ulcer, esophagitis, gastritis or hiatus hernia
* family history of thalassemia, sickle cell anemia, or malabsorption syndrome
* hypersensitivity to iron preparations or current use of iron supplementation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | At 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. MRCOG. PhD, Study Chair — Faculty of Medicine, Mansoura University; Ahmed Ismail, MBBCh, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Kamdi SP, Palkar PJ. Efficacy and safety of ferrous asparto glycinate in the management of iron deficiency anaemia in pregnant women. J Obstet Gynaecol. 2015 Jan;35(1):4-8. doi: 10.3109/01443615.2014.930098. Epub 2014 Jun 24. PMID 24959663